CLINICAL TRIAL: NCT05447221
Title: Automatic Evaluation of the Severity of Gastric Intestinal Metaplasia With Pathology Artificial Intelligence Diagnosis System: a Diagnostic Test
Brief Title: Automatic Evaluation of the Severity of Gastric Intestinal Metaplasia With Pathology Artificial Intelligence Diagnosis System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice President of Qilu Hospital, Shandong University
Other Study IDs: 2022-SDU-QILU-110
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Gastric Intestinal Metaplasia; Artificial Intelligence; Pathology; Gastric Cancer
Keywords: gastric cancer; Gastric Intestinal Metaplasia; Digital Pathology; Whole Slide Image
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsies from the gastric antrum and body will be prospectively collected and prepared as whole slide images for histology examination and model validation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Whole slide images of gastric biopsy specimens: Whole slide images of gastric biopsy specimens
  Interventions: Diagnostic Test: The diagnosis of Artificial Intelligence and pathologists

INTERVENTIONS:
Diagnostic Test: The diagnosis of Artificial Intelligence and pathologists — Pathologists and AI will assess the severity of intestinal metaplasia and judge the tumor area of whole slide images of gastric biopsy specimens independently. In addition, the pathologists can not see the diagnosis of AI.

SUMMARY:
The OLGIM staging system is highly recommended for a comprehensive assessment of GIM severity to evaluate patients' gastric cancer risk. However, its need to take at least 4 biopsies is not clinically feasible due to a serious shortage of pathologists compared with the large number of gastric cancer screening population.

We plan to develop a Digital Pathology artificial intelligence diagnosis system (DPAIDS), to automatically identify tumor areas in whole slide images(WSI) and quickly and accurately quantify the severity of intestinal metaplasia according to the proportion of intestinal metaplasia areas.

DETAILED DESCRIPTION:
Gastric cancer is the fifth most prevalent malignancy and the third most deadly worldwide, and intestinal metaplasia (IM) is a common precancerous state that is closely associated with gastric carcinogenesis .The OLGIM staging system is highly recommended for a comprehensive assessment of GIM severity to evaluate patients' gastric cancer risk. However, its need to take at least four biopsies is not clinically feasible due to a serious shortage of pathologists compared with the large number of gastric cancer screening population. Developing automated screening methods can reduce the heavy diagnostic workload. With advances in digital pathology scanning devices and deep learning technologies, whole-slide images (WSI) have been used to develop automated cancer diagnostic systems.

We plan to develop a Digital Pathology artificial intelligence diagnosis system (DPAIDS), to automatically identify tumor areas in whole slide images(WSI) and quickly and accurately quantify the severity of intestinal metaplasia according to the proportion of intestinal metaplasia areas. Then biopsies will be prospectively collected and prepared as WSI for model validation.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 40-75 years who undergo the gastroscopy examination and biopsy

Exclusion Criteria:

* patients with severe cardiac, cerebral, pulmonary or renal dysfunction or psychiatric disorders who cannot participate in gastroscopy
* patients with previous surgical procedures on the stomach
* patients with contraindications to biopsy
* patients who refuse to sign the informed consent form

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who receive the gastrointestinal endoscopy examination and screened that fulfill the eligibility criteria at Qilu Hospital, Shandong University will be enrolled into the study
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic performance of AI model to assess the severity of intestinal metaplasia | 2 years
  The diagnostic performance of AI model to assess the severity of intestinal metaplasia in a single biopsy tissue slide: Accuracy, sensitivity, and specificity

SECONDARY OUTCOMES:
Accuracy of the digital pathological AI model to identify tumor regions | 2 years
  Accuracy of the digital pathological AI model in identifying tumor regions in the whole slide images
Accuracy of digital pathological AI models to identify glands, mucosal epithelium, and intestinal metaplasia in non-neoplastic areas | 2 years
  Accuracy of digital pathological AI models to identify glands, mucosal epithelium, and intestinal metaplasia in non-neoplastic areas

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD, PhD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China